CLINICAL TRIAL: NCT04242550
Title: Executive Function Training for Binge Eating Disorder and Comorbid Mood/Anxiety Disorders
Brief Title: Binge Eating Anxiety and Mood
Acronym: BEAM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: Brain & Behavior Research Foundation (Other)
Responsible Party: Principal Investigator, Dawn Eichen, Assistant Adjunct Professor, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NARSAD YI 27943
Record Dates: First submitted 2020-01-23; First posted 2020-01-27 (Actual); Last update posted 2022-06-06 (Actual); Status verified 2022-06

CONDITIONS: Binge-Eating Disorder; Binge Eating; Anxiety Disorders; Mood Disorders
MeSH Terms: conditions — Binge-Eating Disorder; Bulimia; Anxiety Disorders; Mood Disorders | interventions — Beds; Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Executive Function- Enhanced CBT for BED (EF-BED+CBT) (Experimental): EF-BED+CBT will combine CBT with executive function training, enhancing CBT with a focus on teaching compensatory strategies, habit learning, and plan for generalization to real-world behaviors.
  Interventions: Behavioral: Executive Function- Enhanced CBT for BED (EF-BED+CBT); Behavioral: Cognitive Behavioral Therapy (CBT)
- Cognitive Behavioral Therapy (CBT) (Active Comparator): CBT will be based on the "Overcoming Binge Eating" book. CBT addresses disturbed eating patterns and problematic thoughts/beliefs related to eating, shape and weight that contribute to binge eating. CBT is the current gold standard treatment for BED.
  Interventions: Behavioral: Cognitive Behavioral Therapy (CBT)

INTERVENTIONS:
Behavioral: Executive Function- Enhanced CBT for BED (EF-BED+CBT) — EF-BED+CBT will combine CBT (see description below) with executive function training. EF-BED will focus on teaching compensatory strategies to enhance adherence to the strategies recommended in CBT.
  Arms: Executive Function- Enhanced CBT for BED (EF-BED+CBT)
Behavioral: Cognitive Behavioral Therapy (CBT) — CBT will be based on the "Overcoming Binge Eating" book. All participants will be provided a copy of the book. CBT addresses disturbed eating patterns and problematic thoughts/beliefs related to eating, shape and weight that contribute to binge eating. CBT is the current gold standard treatment for BED.

SUMMARY:
Binge Eating Disorder (BED) is the most common eating disorder, and currently, the best behavioral treatments only work for 40-60% of adults. BED often co-occurs with mood and anxiety disorders, and both are associated with neurocognitive deficits related to executive function (EF). These EF deficits contribute to worsening BED symptoms and make it difficult for these adults to adhere to treatment recommendations. The proposed study aims to develop an EF training enhanced behavioral treatment for BED and compare its effectiveness to the standard cognitive behavioral therapy for patients with BED and a co-occurring mood or anxiety disorder.

DETAILED DESCRIPTION:
A randomized controlled trial (RCT) will evaluate an EF training enhanced cognitive behavioral therapy (CBT) for BED (EF-BED+CBT) compared to standard CBT in patients with BED and a comorbid mood/anxiety disorder to assess the feasibility, acceptability, and preliminary efficacy of EF-BED+CBT in reducing binge eating, impairment, and comorbid depression/anxiety symptoms. Adult participants with BED and comorbid mood/anxiety disorder will be randomized to a four month remote treatment of either EF-BED+CBT or CBT alone. Participants will be assessed at baseline, following treatment (month 4) and 2-month follow-up (month 6).

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65
* Ability to read English at a 6th grade level
* Clinical or subclinical BED and at least one comorbid mood or anxiety disorder

Exclusion Criteria:

* Known cognitive disability (e.g., brain injury with loss of consciousness >30 min, intellectual disability)
* Psychosis
* Psychiatric condition that could interfere with program participation (e.g., substance abuse, suicide attempt within previous 6 months, active purging, active suicidality)
* Currently pregnant, lactating or plan to be in the timespan of program follow-up
* Change in psychotropic medication or other medication that could have impact on weight, binge eating or anxiety/mood symptoms during the previous 3 months
* Participating in an organized program for overeating

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2020-06-23 (Actual); Primary Completion 2021-11-24 (Actual); Study Completion 2021-11-24 (Actual)

PRIMARY OUTCOMES:
Feasibility as measured by number of treatment sessions attended | Over the course of 4 months of treatment
  Attendance at Treatment Sessions
Acceptability | At 4 months
  Ratings of usefulness of treatment measured by responses to Likert-type ratings developed by the study team.

SECONDARY OUTCOMES:
Binge Eating | Through study completion, an average of 6 months
  Change in binge eating episodes measured by the Eating Disorder Examination interview
Impairment | Through study completion, an average of 6 months
  Change in impairment measured by the Clinical Impairment Assessment (CIA). The CIA is a 16-item questionnaire with possible scores ranging from 0-48 with a higher score indicating a greater level of impairment.

OTHER OUTCOMES:
Anxiety Symptoms | Through study completion, an average of 6 months
  Change in anxiety symptoms measured by the General Anxiety Disorder-7 (GAD-7). The GAD-7 is a 7-item questionnaire with scores ranging from 0-21 and a higher score indicating greater anxiety severity.
Depression Symptoms | Through study completion, an average of 6 months
  Change in depression symptoms measured by the Patient Health Questionnaire-9 (PHQ-9). The PHQ-9 is a 9-item questionnaire with scores ranging from 0-27 and a higher score indicating greater depression severity.

CONTACTS AND LOCATIONS:
Overall Officials: Dawn M Eichen, PhD, Principal Investigator — UC San Diego
Locations (1):
- Ucsd Chear, San Diego, California, United States

REFERENCES:
- [Derived] Eichen DM, Strong DR, Twamley EW, Boutelle KN. Adding executive function training to cognitive behavioral therapy for binge eating disorder: A pilot randomized controlled trial. Eat Behav. 2023 Dec;51:101806. doi: 10.1016/j.eatbeh.2023.101806. Epub 2023 Aug 29. PMID 37660487